CLINICAL TRIAL: NCT04069429
Title: Radiation Dose in Humans From Orally Administered Tc99m-Heparin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Gerald J. Gleich, Principal Investigator, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB_00058734
Record Dates: First submitted 2019-07-27; First posted 2019-08-28 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Technetium; Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: dose assessment of orally administration of Tc99m-Heparin in healthy control and Eosinophilic Esophagitis patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Controls (Experimental): 7 controls (subjects without GI symptoms and known GI disease), subjects will receive the radiopharmaceutical agent orally
  Interventions: Radiation: Computerized Tomography scan; Radiation: Single Photon Emission Computed Tomography scans; Drug: Technetium Tc 99M; Radiation: Planar Images; Procedure: Esophagogastroduodenoscopy
- Eosinophilic Esophagitis Patients (Experimental): 10 patients with diagnosed EoE (greater than 15 eosinophils per HPF) on esophageal biopsy will be included as the diseased population, subjects will receive the radiopharmaceutical agent orally
  Interventions: Radiation: Computerized Tomography scan; Radiation: Single Photon Emission Computed Tomography scans; Drug: Technetium Tc 99M; Radiation: Planar Images; Procedure: Esophagogastroduodenoscopy

INTERVENTIONS:
Radiation: Computerized Tomography scan — imaging scan from a person's eyes to their thighs
  Other Names: CT scan
Radiation: Single Photon Emission Computed Tomography scans — imaging scan taken during, and after, the administration of the radioactive agent
  Other Names: SPECT scans
Drug: Technetium Tc 99M — subjects are administered radioactive heparin as part of study participation.
  Other Names: Radioactive Heparin
Radiation: Planar Images — 2 dimensional imaging - whole body planar scans
Procedure: Esophagogastroduodenoscopy — esophagogastroduodenoscopy with tissue biopsies

SUMMARY:
This is a research study of a new agent used for evaluation of inflammation in the GI tract. This agent is investigational and thus is being studied to determine appropriate dosing and administration in both normal controls (i.e. people without gastrointestinal complaints) and patients with eosinophilic disease (i.e. those with an immune reaction and inflammation in their bodies with a certain cell called an eosinophil).

The study will test whether the radiolabeled agent will bind to the inflammation of eosinophilic esophagitis patients because an animal model of eosinophilic esophagitis which shows the striking deposition of eosinophil granule proteins is not available.

ELIGIBILITY:
Inclusion Criteria:

* 10 patients with diagnosed EoE (greater than 20 eosinophils per HPF) on esophageal biopsy will be included as the diseased population
* 7 controls (subjects without GI symptoms and known GI disease)

Exclusion Criteria:

* bleeding diathesis or contraindication to esophageal biopsies
* severe sleep apnea
* incarceration
* pregnancy
* inability to lie flat for 2 hours
* history of bleeding disorder
* Use of steroids
* Breast feeding
* Allergy to heparin or history of severe reaction to heparin
* allergy to mucomyst or severe asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Biodistribution of Tc99m-heparin | over approximately 24-26 hours
  Biodistribution of Tc99m-heparin to the esophagus and other organs, especially of the gastrointestinal tract as judged by planar scans and by single photon emission computed tomography scans.
Calculation of organ doses | over approximately 24-26 hours
  Calculation of organ doses from the oral administration of Tc99m-heparin. The organ doses will be measured in miliSieverts using a computer program called OLINDA (Version 2).

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gleich, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No